CLINICAL TRIAL: NCT03046966
Title: Manikin To Patient Intubation: Does It Translate?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 205053
Record Dates: First submitted 2017-02-02; First posted 2017-02-08 (Estimated); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-04

CONDITIONS: Intubation; Difficult or Failed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Control: No Training (Other): Does not receive hands-on intubation training in the Simulation Lab.
  Interventions: Other: Intervention: Control No Training
- Intervention: Receives Training (Other): Receives hands-on intubation training in the Simulation Lab.
  Interventions: Procedure: Intervention: Receives Training

INTERVENTIONS:
Procedure: Intervention: Receives Training — • Complete a Hands-on Intubation in the Simulation Lab with PI instructing:
  * Using state of the art technology, a Storz C-MAC video laryngoscope
  * Identifying anatomical landmarks
  * Practice on the manikin until intubation occurs within 15 seconds
  Arms: Intervention: Receives Training
Other: Intervention: Control No Training — • Does not receive simulation training with PI. Only standard training.
  Arms: Intervention Control: No Training

SUMMARY:
This study evaluates a new approach to the instruction of pediatric residents in the skill of neonatal intubation. Half of the participants will receive focused simulation training and cognitive instruction while the other half will not. The collected data from both groups will be compared.

DETAILED DESCRIPTION:
Current findings suggest that the training of pediatric residents is not sufficient prior to "live" tracheal intubations in the critical care setting. The current one to two days of airway management training as a part of resuscitation training (such as Pediatric Advanced Life Support (PALS) or Neonatal Resuscitation Program (NRP) is not sufficient to provide safe intubation skills.

This study will develop and implement tracheal intubation training using concepts of deliberate practice modeled after Ericsson. The concepts include focused training on a specific task, immediate feedback, time for problem solving and evaluation, and opportunities for repeated performance using a manikin. This proposal is an attempt to develop such a training model. Video recordings of live intubations will be reviewed and evaluated. The data between the two groups will be compared to see if there is improved intubation skills of live patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female residents from 18-89 years of age who have been assigned to the Neonatal Intensive Care Unit (NICU) for a monthly rotation are eligible to participate. At the beginning of all NICU rotations, all pediatric residents will be invited to participate in this research.

Exclusion Criteria:

* Any pediatric resident who does not wish to participate

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Hall, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rumpel J, O'Neal L, Kaukis N, Rogers S, Stack J, Hollenberg J, Hall RW. Manikin to patient intubation: does it translate? J Perinatol. 2023 Feb;43(2):233-235. doi: 10.1038/s41372-022-01553-9. Epub 2022 Nov 11. No abstract available. PMID 36369530

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 102 residents were approached for enrollment. 102 residents were consented and randomized to intervention or control based on month of NICU rotation.
Groups:
- Intervention: Receives Training: Receives hands-on intubation training in the Simulation Lab.
  Intervention: Receives Training: • Complete a Hands-on Intubation in the Simulation Lab with PI instructing:
  * Using state of the art technology, a Storz C-MAC video laryngoscope
  * Identifying anatomical landmarks
  * Practice on the manikin until intubation occurs within 15 seconds
Period: Overall Study
Arm/Group | Intervention Control: No Training | Intervention: Receives Training
Started | 51 | 51
Completed | 51 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group: Control: No Training Residents received standard training consisting of intern orientation.
- Intervention Group: Intervention Group: Received individualized with a neonatologist at the beginning of the NICU rotation utilizing video laryngoscope and a neonatal mannequin. These residents also received standard training at intern orientation.
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 51 | 102
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 48 | 48 | 96
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51 | 51 | 102
Level of Training (year) [Count of Participants; unit: Participants]
  First year | 30 | 36 | 66
  Second year | 14 | 5 | 19
  Third year | 7 | 8 | 15
  Fourth Year | 0 | 2 | 2
Comfort with Intubation [Count of Participants; unit: Participants]
  Not very comfortable | 22 | 24 | 46
  Somewhat comfortable | 12 | 10 | 22
  Neutral | 9 | 7 | 16
  Comfortable | 8 | 10 | 18
  Very comfortable | 0 | 0 | 0
Baseline Successful Intubation Rate [Count of Participants; unit: Participants]
  0-25% | 9 | 9 | 18
  25-50% | 6 | 3 | 9
  50-75% | 12 | 8 | 20
  75-100% | 6 | 9 | 15
  Not Applicable | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Successful Intubation Encounters on Live Neonates
Description: Residents reported the number of successful intubation encounters they performed during their one month long NICU rotation. A successful intubation encounter is an intubation procedure where the resident successfully placed the the endotracheal tube (ETT) through the vocal cords into the trachea. Placement was confirmed with xray, chest auscultation, improvement in heart rate, and CO2 detectors.
Time Frame: 1 month- neonatal intensive care unit (NICU) rotation
Measure: Mean (Standard Error); unit: Successful Intubation Encounters
Units Other Than Participants: Intubation Encounters
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 51 | 51
Number analyzed (Intubation Encounters) | 93 | 119
Successful Intubation Encounters | 1.02 (0.167) | 1.18 (0.183)

2. Secondary Outcome: Successful Intubations on the First Attempt
Description: Each resident reported the number of successful intubation encounters requiring one attempt on live infants during their NICU rotation. An intubation attempt occurs any time the laryngoscope enters the neonate's mouth. There can be multiple intubation attempts in one intubation encounter. However this outcome focuses on intubation encounters where the neonate was intubated on the first attempt by the resident.
Time Frame: 1 month- NICU rotation
Population: Six residents in the Control group did not report the number of successful intubation encounters completed with only one attempt.
Measure: Mean (Standard Error); unit: Successful First Attempt Intubations
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 45 | 51
Successful First Attempt Intubations | 0.578 (0.133) | 0.840 (0.161)

3. Secondary Outcome: Total Number of Intubation Encounters Performed by Each Resident During Their NICU Rotation
Description: The mean number of intubation encounters performed by each resident during their NICU rotation was compared between the Control and Intervention groups.
Time Frame: 1 month- NICU rotation
Measure: Mean (Standard Error); unit: Intubation Encounters
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 51 | 51
Intubation Encounters | 1.82 (0.189) | 2.33 (0.214)

4. Secondary Outcome: Change in Time to Intubate the Mannequin
Description: All study residents intubated the mannequin before and after their NICU rotation. The total time of the mannequin intubation encounter was recorded. The difference in the time from end of the NICU rotation and the baseline time (beginning of the NICU rotation) was calculated.
Time Frame: 1 month- NICU rotation
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 51 | 51
Seconds | 18.6 (9.61) | 37.6 (8.7)

ADVERSE EVENTS:
Time Frame: NICU rotation (1 month)
Arm/Group | Intervention Control: No Training | Intervention: Receives Training
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 0/51 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT03046966/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT03046966/SAP_001.pdf